CLINICAL TRIAL: NCT04411277
Title: Time in Range (TIR) and Time Below Range (TBR) in Insulin-Treated Elderly Patients With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Cline Research Center (Other)
Collaborators: Abbott Diabetes Care (Industry)
Responsible Party: Principal Investigator, Silmara Leite, Director, Cline Research Center
Other Study IDs: ADC-OUS-IIS-19-47
Record Dates: First submitted 2020-05-06; First posted 2020-06-02 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Continuous Glucose Monitoring
Keywords: Type 2 Diabetes; Elderly; Continuous Glucose Monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- T2DM Elderly on Insulin CGM: 70 patients with type 2 diabetes > 65 years of age taking insulin as treatment. The sample size was calculated to estimate the minimal number of patients necessary to describe the mean TIR (minutes/day).
  Interventions: Device: Application of the FreeStyle Libre Flash Glucose CGM.; Diagnostic Test: InBody 270 multifrequency bioimpedance

INTERVENTIONS:
Device: Application of the FreeStyle Libre Flash Glucose CGM. — Assessment of glycemic control and hypoglycemia, adherence to therapy and CGM use.
Diagnostic Test: InBody 270 multifrequency bioimpedance — analysis of body composition to calculate appendicular skeletal muscle.

SUMMARY:
Prospective observational cohort study. Elderly patients >65 years with type 2 diabetes mellitus (T2DM) on insulin therapy and HbA1c between 7% and 9%, with or without oral agents, will be identified from medical records and invited to participate. Patients will wear a FreeStyle Libre Flash CGM during a 6-week study period.

Using CGM technology, we will assess an efficacy outcome : time in range (TIR) between 70-180 mg/dl and a safety outcome: incidence of hypoglycemia (time below range (TBR) less than 70, 54, and 40 mg/dl in insulin treated older adults with T2DM.

Patients will return to clinic every 2 weeks for new continuous glucose monitoring (CGM) placement, assessment of glycemic control and hypoglycemia, adherence to therapy and CGM use.

CGM data will be downloaded every 2 weeks.

DETAILED DESCRIPTION:
Prospective observational cohort study. Patients over 65 years of age, with TDM2 using insulin with or without the use of associated oral antidiabetic agents and with HbA1c between 7% and 9%, will be identified by medical records at the Hospital da Cruz Vermelha Brasileira-Filial do Paraná and they will be invited to participate in the study by telephone and forwarded to the research center Cline Research Center where the study procedures will be carried out. Patients from the private clinic of neurology and endocrinology Cline will also be invited by telephone. In this way the sample of patients will include patients from the public and private health system.

On the first visit to the research centers, after signing the informed consent form (ICF), patients will be evaluated for the presence of other comorbidities associated with diabetes such as the presence of cardiovascular disease, hypertension and dyslipidemia.

The screening for the presence of sarcopenia will be performed with the application of the SARC-F questionnaire; measuring muscle strength with grip strength; the functional test of getting up from the chair without supporting the arms and walking for 3 meters, turning 180º and returning to sit. The time in which the elderly person performs this task is timed and the time up to 20 seconds is considered normal.

Patients will undergo a complete physical examination and body composition analysis using the InBody 270 multifrequency bioimpedance to calculate the appendicular skeletal musculature.

After the first evaluation at the research centers, patients will be referred to partner laboratories that use the same methodologies for measuring HbA1c, blood count, urea, creatinine, glutamic oxalacetic transaminase (TGO) and glutamic-pyruvic transaminase (TGP), which will be performed only at the initial visit.

During the second visit to the research center, the FreeStyle Libre Flash interstitial glucose sensor will be inserted for the first time in the posterior and upper arm and the patient will be instructed to read the glucose at least 10 times a day, being sure to check glucose for a period longer than 8 hours. The patient should be instructed to return to the research center every 2 weeks to change the sensor until completing the 6-week period.

The patient's travel to the research center will be reimbursed by the study team. The study will be carried out at the Hospital da Cruz Vermelha Brasileira-Filial do Paraná, located in Curitiba in partnership with the independent research center Cline Research Center (CRC). Eligible patients will be randomly selected from clinical outpatients at participating institutions, concomitantly.

ELIGIBILITY:
Inclusion Criteria:

* Age > 65 years
* Known history of type 2 Diabetes Mellitus
* BMI between 18.5 and 35kg/m2
* HbA1c between 7% and 9.0%
* Insulin with or without oral agent treatment for diabetes mellitus

Exclusion Criteria:

* Patients using GLP1 (Glucagon-like peptide-1) agonists
* Patients with eGFR<30 (epidermal growth factor receptor) using (calculated CKD EPI)
* Anemia (Hb<11 grams)
* Chronic liver chronic disease (ALT>3xULN)
* Use of glucocorticoids within 3 months preceding the investigation
* Neoplasia treatment
* Inability by the patient or caretaker to commit to protocol instructions and visit schedule.
* Type 1 diabetes

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients >65 years with T2DM on insulin therapy and HbA1c between 7% and 9%, with or without oral agents, will be identified from medical records and invited to participate. Patients will wear a FreeStyle Libre Flash CGM during a 6-week study period.
Sampling Method: Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Primary outcome is time in range (TIR) | 04-07-2021
  TIR between 70-180 mg/dL in insulin treated in patients older than 65 years.

SECONDARY OUTCOMES:
-Frequency of hypoglycemia (<70mg/dL, <54mg/dL) to measure Time Bellow Range | 04-07-2021
  * percentage of patients with greater than 5%-time below glucose target (<70 mg/dL);
  * diurnal and nocturnal hypoglycemia;
-Time in hyperglycemia > 180, 250 mg/dL to measure Time Above Range | 04-07-2021
  * percentage of patients with greater than 5%-time glucose above 250mg/dL
  * percentage of patients with greater than 25%-time glucose above 180mg/dL
-Adherence to CGM use and sensor utilization for diabetes care management using CGM | 04-07-2021
  -assessing the percentage of captured sensor data
- Rate of emergency room visits and hospitalization | 04-07-2021
  -changing insulin type and dose to prevent hospitalization
-Glucose Variability | 04-07-2021
  * glycemic variability standard deviation and MAGE(mean amplitude of glycemic excursions)
  * glucose variability will be calculated as % coefficient of variation %CV= (standard deviation (SD)/mean glucose x 100%)

CONTACTS AND LOCATIONS:
Overall Officials: Silmara Leite, MD, PhD, Principal Investigator — Cline Research Center
Locations (1):
- Cline Research Center, Curitiba, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The physiology of endocrine systems with ageing — http://www.ncbi.nlm.nih.gov/pubmed/30017799
- See also: Diabetes in the older patient: heterogeneity requires individualization of therapeutic strategies — https://www.ncbi.nlm.nih.gov/pubmed/29417185
- See also: Continuous Glucose Monitoring Versus Usual Care in Patients With Type 2 Diabetes Receiving Multiple Daily Insulin Injections: A Randomized Trial. — https://www.ncbi.nlm.nih.gov/pubmed/28828487
- See also: Estimating the mean and variance from the median, range, and the size of a sample. — https://www.ncbi.nlm.nih.gov/pubmed/15840177
- See also: A power primer. — https://www.ncbi.nlm.nih.gov/pubmed/19565683
- See also: The Relationship of Hemoglobin A1C to Time-in-Range in Patients with Diabetes. — https://www.ncbi.nlm.nih.gov/pubmed/30575414